CLINICAL TRIAL: NCT03796429
Title: A Single-arm, Single-center, Prospective Clinical Study of the Efficacy and Safety of Chemotherapy Combined With Toripalimab in the Treatment of Advanced Biliary Tract Cancer
Brief Title: A Study of the Efficacy and Safety of Chemotherapy Combined With Toripalimab in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other); OrigiMed (Industry)
Responsible Party: Principal Investigator, Tianshu Liu, Head of Medical oncology, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ZS-BC001
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Biliary Tract Cancer
Keywords: Advanced Biliary Tract Cancer; PD-1 antibody(Toripalimab); first-line chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GS+Toripalimab (Experimental)
  Interventions: Drug: GS+Toripalimab

INTERVENTIONS:
Drug: GS+Toripalimab — Patients will be given treatment as below once recruited: PD-1 antibody Toripalimab（240mg, iv, q3w），combined with GS regimen(gemcitabine 1000mg／m2 ，d1,d8 + S1 40-60mg bid*14d，Q21d).
  The treatment will be continued until emerging of disease progression or intolerable adverse effects (The upper time limit for treatment is 2 years).

SUMMARY:
1. Target population: patients with advanced biliary tract cancer (including gallbladder carcinoma, intrahepatic and extrahepatic cholangiocarcinoma) .
2. Primary objective: progression free survival (PFS)/ overall survival (OS) of first-line chemotherapy plus PD-1 antibody (Toripalimab) in patients with advanced biliary tract cancer.

Secondary objectives:

1. objective response rate (ORR) of first-line chemotherapy plus PD-1 antibody (Toripalimab)
2. safety of first-line chemotherapy plus PD-1 antibody (Toripalimab)

3.Trial design: This is a monocenter, single arm, phase II study to evaluate the efficacy and safety of first-line chemotherapy plus PD-1 antibody (Toripalimab) in patients with advanced advanced biliary tract cancer.

4.Treatment plan: Patients will be given treatment as below once recruited: PD-1 antibody Toripalimab（240mg, iv, q3w），combined with GS regimen(gemcitabine 1000mg／m2 ，d1,d8 + S1 40-60mg bid*14d，Q21d).

The treatment will be continued until emerging of disease progression or intolerable adverse effects (The upper time limit for treatment is 2 years).

5.Number of subjects: 40 patients. Number of centers: 1 sites ( Fudan University Affiliated Zhongshan Hospital).

DETAILED DESCRIPTION:
Backgrounds:

Toripalimab (JS-001) is a PD-1 antibody developed by Shanghai Jun Shi Biomedical technology Co. Ltd. Nowadays, eighteen clinical trials of this drug have been conducted in patients with different types of advanced malignant tumor. Until now, Toripalimab has exhibited favorable safety in recruited patients. Incidence rate of SAE is 14.7%. JS001-Ib-CRP-1.0 is a phase Ib/II basket trial, aiming at evaluating safety and efficacy of JS001 in treating advanced gastric adenocarcinoma, esophageal squamous cell carcinoma, nasopharyngeal carcinoma and head and neck squamous cell carcinoma.The interim analyses results of 161 patients show that the ORR is 22.4%.

Now, the standard chemotherapies regimen for advanced biliary tract cancer include gemcitabine, platinum and fluorouracil; Considering the synergistic effect of chemotherapy and immune therapy, the investigators choose GS regimen (gemcitabine+S1) to combine Toripalimab.

the investigators will shut down the study in advance, if unpredicted SAE or low efficacy occur.

Patients with abnormal autoimmune status, unfavorable body function, factors impeding drug taking, absorption and metabolism will be excluded. Study participants with disease progression or severe/ intolerant toxicity during treatment will withdraw the study.

Hyper-progressive disease is defined as 1) progression 2) more than doubled growth rate 3) tumor volume increase >50% in 2 months after initialing the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female. Age ≥ 18 years and ≤75 years.
2. histologically documented advanced biliary duct cancer, including gallbladder cancer, intrahepatic and extrahepatic cholangiocarcinoma, specimen within a year available for test (at least 10 pathological sections) .
3. at least one measurable lesion in abdominal CT/MRI according to RESIST 1.1 is required.
4. Karnofsky score≥ 80.
5. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥90g/L.
6. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.
7. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 60 ml/min.
8. Adequate coagulation function: INR/PT≤ 1.5 x ULN, aPTT≤ 1.5 x ULN.
9. No serious concomitant disease that will threaten the survival of patients to less than 5 years.
10. Written (signed) informed consent.
11. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
12. Female patients should not be pregnant or breast feeding.
13. Agree to take contraception measures during treatment and in 120 days after last dose of Toripalimab or in 180 days after last dose of chemo.

Exclusion Criteria:

1. history of chemo, radiation, immune therapy or radical resection for the biliary tract cancer, except those patients who relapsed after 6 months since the last time of adjuvant therapy.
2. patients with active autoimmune disease or history of refractory autoimmune disease.
3. patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured locally tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ.
4. uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment.
5. patients who have digestive tract bleeding in 2 weeks before recruitment or with high risk of bleeding.
6. perforation / fistula of GI tract in 6 months before recruitment.
7. losing over 20% body weight in 2 months before recruitment.
8. pulmonary disease history: interstitial pulmonary disease, non-infective pneumonitis, pulmonary fibrosis, acute pulmonary disease.
9. uncontrollable systemic diseases, including diabetes, hypertension, etc.
10. severe chronic or active infections in need of systemic antibacterial, antifungal, or antiviral treatment, including TB or HIV, etc.
11. patients with untreated chronic hepatitis B or HBV DNA over 500 IU/ml or positive HCV RNA.
12. patients with any cardiovascular risk factors below:

    1. cardiac chest pain occurring in 28 days before recruitment, defined as moderate pain that limits daily activity.
    2. pulmonary embolism with symptoms occurring in 28 days before recruitment.
    3. acute myocardial infarction occurring in 6 months before recruitment.
    4. any history of heart failure reaching grade 3/4 of NYHA in 6 months before recruitment.
    5. ventricular arrhythmias of Grade 2 or grater in 6 months before recruitment, or accompanied by supraventricular tachyarrhythmias requiring medical treatment.
    6. cerebrovascular accident within 6 months before recruitment.
13. patients with peripheral neuropathy NCI CTC AE grade 1, except those with only deep tendon reflex disappearing.
14. moderate or severe renal injury [creatinine clearance rate≤50 ml/min (according to Cockroft & Gault equation)], or Scr>ULN.
15. allergic to any drug in this study.
16. history of allogeneic stem cell transplantation or organ transplantation.
17. use of steroids (dosage>10mg/d prednisone) or other systemic immune suppressive therapy in 14 days before recruitment, except patients treated with regimens below: a. steroids for hormone replacement (dosage>10mg/d prednisone); b. steroids for local application with little systemic absorption; c. short -term (≤ 7 days) steroids for preventing allergy or vomiting.
18. vaccinated with live vaccine in 4 weeks before recruitment.
19. receiving immune (interleukin, interferon, thymin) treatment or treatment of other trials in 28 days before recruitment.
20. receiving palliative radiation in 14 days before recruitment.
21. history of anti PD-1, PD-L1, PD-L2 or any other specific T cell co-stimulation or checkpoint pathway targeted treatment.
22. receiving operation in 28 days before recruitment, only if the operation is a minimally invasive one e.g. PICC.
23. for patients with uncontrolled epilepsy, CNS diseases or history of mental disorder, researchers should evaluate whether their diseases will impede their signing of informed consent or compliance of treatment.
24. existing of potential situation which will impede drug administration or affect toxicity analysis or alcohol/ drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) of GS regimen plus PD-1 antibody (Toripalimab) | 36 months after the last subject participating in
  PFS is defined as time interval from recruitment to tumor progression or censoring. Tumor progression is defined as below: 1) relapse of primary lesion 2) emerging of new lesion 3) distant metastasis 4) death of any reason 5)tumor progression according to RESIST 1.1 on CT/MRI.
overall survival (OS) of GS regimen plus PD-1 antibody (Toripalimab) | 36 months after the last subject participating in
  OS is defined as time interval from recruitment to all-caused death or censoring.

SECONDARY OUTCOMES:
objective response rate (ORR) of GS regimen plus PD-1 antibody (Toripalimab) | 36 months after the last subject participating in
  rate of patients with complete remission (CR) or partial remission (PR) based on RESIST1.1. ORR was evaluated by chest, abdominal & pelvic CT/MRI. Evaluation will be conducted every 6 weeks during treatment, and every 0.5 year after all treatments.
Incidence of adverse Events of GS regimen plus PD-1 antibody (Toripalimab) | 1 month after the last date of treatment
  Adverse events (AE) of chemotherapy will be graded and documented according to NCI-CTC AE v4.03 from the beginning of treatment to 1 months after the last date of treatment. Documentary will include severity, lasting period and occurrence time. Main AEs include vomiting, diarrhea, anemia, leukopenia, thrombocytopenia, hand-foot syndrome, immune related adverse events (including interstitial lung disease, AST/ALT elevations, hypothyroidism and hyperthyroidism,etc) and hyper-progressive tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China